CLINICAL TRIAL: NCT06944704
Title: Clinical Study Evaluating Efficacy, Safety and Molecular Mechanism of Pentoxifylline Supplementation in Patients With Hepatic and Post Hepatic Jaundice
Brief Title: Evaluation of Efficacy, Safety and Molecular Mechanism of Pentoxifylline Supplementation in Patients With Hepatic and Obstructive Jaundice
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Samah Hussein Mohamed, Principal investigator, M.Sc. in Clinical Pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP/RE1/24Ph-1
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-01

CONDITIONS: Hepatobiliary Disorders
Keywords: Jaundice; Pentoxifylline; TAC; TNF-α; Bilirubin
MeSH Terms: conditions — Digestive System Diseases; Jaundice | interventions — Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): 20 patients who will receive supportive treatment for jaundice only, for 3 months.
- PTX arm (Experimental): 20 patients who will receive oral Pentoxifylline 400 mg twice daily in addition to supportive treatment, for 3 months.
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline — Patients will receive oral Pentoxifylline 400 mg twice daily in addition to supportive treatment, for 3 months.
  Arms: PTX arm

SUMMARY:
Investigating the efficacy, safety, and molecular mechanism of Pentoxifylline supplementation in improving elevated direct bilirubin level and liver function tests in patients with hepatic and post-hepatic jaundice

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-70 years old.
* Patients diagnosed with jaundice and increased level direct bilirubin ≥ 3 mg/dL.

Exclusion Criteria:

* Pregnancy.

  * Nursing mothers.
  * Patients with increased indirect bilirubin level.
  * Patients who have Gilbert syndrome or Crigler Najjar syndrome.
  * Patients with Child Paugh C score (10-15 point).
  * History of intolerance and hypersensitivity to Pentoxifylline or to xanthine derivatives such as caffeine, theophylline.
  * Recent hemorrhage.
  * Patients who have risk factors potentially complicated by hemorrhage.
  * Taking anticoagulants or antiplatelet therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Change in total antioxidant capacity (TAC) level, | The participants will be assessed before initiation of the study (baseline), and at the end of the study up to 12 weeks.
  Assessment of total antioxidant capacity (TAC) level by ELISA Kits according to manufacturer's instructions.
Change in tumor necrosis factor alpha (TNF-α) | The participants will be assessed before initiation of the study (baseline), and at the end of the study up to 12 weeks.
  Assessment of tumor necrosis factor alpha (TNF-α) level by ELISA Kits according to manufacturer's instructions.

SECONDARY OUTCOMES:
Follow up of liver function | The participants will be assessed before initiation of the study (baseline), and at the end of the study up to12 weeks.
  measurement of alanine transaminase (ALT) and aspartate transaminase (AST) both in U/L from blood samples will be assessed for all participants.
Adverse events and toxicity | up to 12 weeks
  Adverse events and toxicity will be graded using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided